CLINICAL TRIAL: NCT00641225
Title: An Ascending Single Dose Study Of The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of SBI-087 Administered To Subjects With Rheumatoid Arthritis
Brief Title: Study Evaluating Single Doses Of SBI-087 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3227K1-1000; B2261001
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Ascending Single Dose; Safety; Pharmacokinetics; Open-label
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — SBI-087

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SBI-087
  Interventions: Drug: SBI-087

INTERVENTIONS:
Drug: SBI-087 — Single IV doses of SBI-087 from 0.015 mg/kg to 2 mg/kg and Single SC doses of SBI-087 from 50 mg to 300 mg.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of single doses of SBI-087 in subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Man or nonlactating and nonpregnant woman, aged 18 to 70 years, inclusive, at the screening visit.
* Must meet criteria for rheumatoid arthritis with functional class I to III.
* Diagnosis of rheumatoid arthritis more than 6 months before study day 1 and rheumatoid arthritis onset after 16 years of age

Exclusion Criteria:

* Any significant health problems other than rheumatoid arthritis.
* Treatment of greater than 10 mg of prednisone per day.
* Treatment with cyclophosphamide.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2011-03-31 (Actual); Study Completion 2011-03-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ascending single doses of SBI-087 in subjects with rheumatoid arthritis. | 12 months

SECONDARY OUTCOMES:
To provide the initial pharmacokinetics and pharmacodynamic profile of SBI-087 in subjects with rheumatoid arthritis. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (3):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Dallas, Texas
- Canada (3):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec

REFERENCES:
- [Derived] Cohen S, Clowse M, Pardo P, Bhattacharya I, Menon S, Gourley I, Diehl A. Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of SBI-087, a CD20-Directed B-cell Depleting Agent: Phase 1 Dose Escalating Studies in Patients With Either Mild Rheumatoid Arthritis or Systemic Lupus. Clin Ther. 2016 Jun;38(6):1417-1434.e2. doi: 10.1016/j.clinthera.2016.03.028. Epub 2016 Apr 21. PMID 27112532
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3227K1-1000&StudyName=Study%20Evaluating%20Single%20Doses%20Of%20SBI-087%20in%20Subjects%20With%20Rheumatoid%20Arthritis